CLINICAL TRIAL: NCT04724395
Title: Prospective Multicenter Cohort Study to Evaluate Disability Following Hospitalization in People of Working-age Surviving COVID-19
Brief Title: Disability Following Hospitalization in People of Working-age Surviving SARS-CoV-2 Infection - COVID-19
Acronym: DisCOVID
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P200601; 2020-A02552-37 (Other: ID-RCB)
Record Dates: First submitted 2020-11-30; First posted 2021-01-26 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2 infection; Post-acute COVID-19; Disability; Health-related quality of life
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Hospitalization — Hospitalization in intensive care and non-intensive care units for COVID-19 followed by usual care

SUMMARY:
The purpose of the study is to describe disability following hospitalization in people of working-age surviving COVID-19.

DETAILED DESCRIPTION:
In December 2019, the Wuhan Municipal Health Committee in China identified an outbreak with viral pneumonia cases of unknown cause. Coronavirus RNA was identified as the causal agent. The disease caused by SARS-CoV-2 has been named COVID-19. While most people with COVID-19 develop uncomplicated illness, approximately 14% develop severe forms of the disease and 5% are critically ill, potentially leaving survivors with non-fatal sequelae. To date, the long-term burden of COVID-19 and patients' perspectives and needs have been left unaddressed. As compared to 2003 SARS outbreak, one can anticipate persisting disability in COVID-19 survivors, including specific post-COVID and non-specific post-intensive care syndromes. The investigators hypothesize that dramatic COVID-19-specific and non-specific mid- and long-term disabilities would persist in people surviving COVID-19.

The main objective will be to provide a deep understanding of non-fatal health outcomes in people surviving COVID-19, by comprehensively and systematically mapping and monitoring, within the WHO ICF framework, disability levels and profiles, in the mid and long terms in people surviving COVID-19.

Disability levels will be assessed at 12 (±7) and 36 (±3) months using:

* Parts 1a (impairments of body functions) and 2 (activity limitation and participation restriction) of the WHO ICF checklist v2.1, administered by a health care provider, and
* Self-administered 36-item WHO Disability Assessment Schedule 2.0 (WHODAS 2.0)

A. The secondary objectives will be to describe COVID-19 specific and non-specific impairments, activity limitations and participation restriction at 12 (±7) and 36 (±3) months in people surviving COVID-19:

* Impairments, participation restrictions and health-related quality of life (HRQoL) at 12 (±7) and 36 (±3) months will be assessed using online specific self-administered questionnaires and face-to-face specific tests.
* Non-pharmacological / pharmacological treatments at baseline, 12 (±7) and 36 (±3) months will be self-reported.
* Total costs, cost drivers and estimated Years-Lived with Disability (YLDs) at 12 (±7) and (36 (±3) months will be calculated.

B. Another secondary objective will be to assess the burden of the patient's SARS-CoV-2 infection on the patient's close relative, between M12-inclusion and M36 patient visits.

• The burden on patient's close relative will be assessed using specific printed self-administered questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adults of working-age (18 to 70 years),
* Hospitalization during the prespecified inclusion period (from March 2020 to March 2021) (NB : in case of transferred patients, inclusion in the DisCOVID study must be carried out in the first place of admission for COVID),
* Laboratory-confirmed SARS-CoV-2 and/or CT-scan showing typical radiological findings,
* SARS-CoV-2 of any duration,
* Ability to comply with study visits,
* Informed written consent

Exclusion Criteria:

* Return home in less than 72 hours
* Absence of health insurance,
* Inability to fluently speak and/or read French language,
* People under tutorship or curatorship and protected adults.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People of working-age surviving COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Post-acute COVID-19 disability from the care provider's perspective, 12 months after hospitalization | At 12 (±7) months after hospitalization
  Disability levels will be assessed using Part 1a (impairments of body functions) and 2 (activity limitation and participation restriction) of the WHO ICF checklist v2.1, administered by a health care provider.
Post-acute COVID-19 disability from the care provider's perspective, 36 months after hospitalization | 36 (±3) months after hospitalization
  Disability levels will be assessed using Part 1a (impairments of body functions) and 2 (activity limitation and participation restriction) of the WHO ICF checklist v2.1, administered by a health care provider
Post-acute COVID-19 disability from the patient's perspectives, 12 months after hospitalization | At 12 (±7) months after hospitalization
  Disability levels will be assessed using the self-administered 36-item WHO Disability Assessment Schedule 2.0 (WHODAS 2.0)
Post-acute COVID-19 disability from the patient's perspectives, 36 months after hospitalization | 36 (±3) months after hospitalization
  Disability levels will be assessed using the self-administered 36-item WHO Disability Assessment Schedule 2.0 (WHODAS 2.0)

SECONDARY OUTCOMES:
Type of treatments | At 12 (±7) and 36 (±3) months after hospitalization
  Non-pharmacological / pharmacological treatments will be self-reported : ER consultations, specialist consultations, laboratory tests, new hospital stay, rehabilitation resource consumption
Acceptable symptom state (questionnaire self-administered on ComPARe IT dedicated platform) | 12(±7) and 36 (±3) months after the first day of the first hospitalization.
  Anchor questions ( 2 questions)
Health-related quality of life (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  EuroQol : ED-5D-5L (5 themes of questions + a scale from 0 to 100, 100 is the best state of health)
Pain (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Brief Pain Inventory (7 scales from 0 to 10 : 10 is the worst pain)
Impairments, activity limitations and participation restrictions, health-related quality of life Fatigue (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Modified Fatigue Impact Scale (8 questions)
Impairments, activity limitations and participation restrictions, health-related quality of life (questionnaires self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Hospital Anxiety and Depression Scale (14 questions with scales from 0 to 3)
Impairments, activity limitations and participation restrictions, health-related quality of life (questionnaires self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Post-Traumatic Stress Disorder Checklist Scale (17 questions with a scale from 1 to 5)
Impairments, activity limitations and participation restrictions, health-related quality of life (questionnaires self-administered on ComPARe IT dedicated platform) | 12 (±7), and 36 (±3) months after the first day of the first hospitalization.
  Brain Injury Complaint Questionnaire (25 questions)
Urinary symptoms, if applicable (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Urinary Symptom Profile (10 questions)
Female sexual dysfunction, if applicable (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Female Sexual Function Index
Erectile dysfunction, if applicable (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  International Index of Erectile Function (5 questions with a scale from 0 to 5)
Global activity limitations and participation restrictions (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  36-Item WHODAS 2.0
Work Ability (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Work Ability Index Single-Item 1 (1 question with a scale from 0 to 10, 10 is the highest ability to work)
Work productivity (questionnaire self-administered on ComPARe IT dedicated platform) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Work Productivity and Activity Impairment questionnaire Single-Item 5 (1 question with a scale from 0 to 10, 10 is the worst productivity)
Comorbidities (score completed by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Charlson comorbidity index (20 items)
Impairments, activity limitations and participation restrictions (checklist completed by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  WHO ICF checklist v2.1
Mobility test to assess the consequences of neurological, cardiorespiratory, osteoarticular or respiratory impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  6 minute walk test
Locomotor impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Timed up and go test
Upper extremities impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Box and Block test
Respiratory impairment (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  MRC Dyspnoea scale
Respiratory impairment (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  NYHA grade
Cognitive impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Montreal Cognitive Assessment
Cognitive impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Frontal Assessment Battery
Muscular impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  MRC-Sum Score
Respiratory impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Sustained Expiration while counting
Muscular impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Grip strength
Muscular impairments (clinical assessment by the investigator during a face-to-face visit) | 12 (±7) and 36 (±3) months after the first day of the first hospitalization.
  Chair rise with arms
Total costs | 12 (±7) and 36 (±3) months after the first day of the first hospitalization
Costs drivers | 12 (±7) and 36 (±3) months after the first day of the first hospitalization
Estimated Years lived with Disability | 12 (±7) and 36 (±3) months after the first day of the first hospitalization
Burden of post-acute COVID-19 on participant's close relative | Between 12 (±7) and 36 (±3) months after the first day of the first hospitalization of the patient.
  Zarit Burden Inventory (22 questions with a scale from 0 to 4) (using printed version of specific self-administered questionnaires completed by the patient' close relative)
Resource utilization | Between 12 (±7) and 36 (±3) months after the first day of the first hospitalization of the patient.
  Resource Utilization in Dementia - Part I (3 items of questions) (using printed version of specific self-administered questionnaires completed by the patient' close relative)
Symptoms of anxiety and/or depression of participant's close relative | Between 12 (±3) and 36 (±3) months after the first day of the first hospitalization of the patient.
  Hospital Anxiety and Depression Scale (using printed version of specific self-administered questionnaires completed by the patient' close relative)
Symptoms of post-traumatic stress | Between 12 (±7) and 36 (±3) months after the first day of the first hospitalization of the patient.
  Post-Traumatic Stress Disorder Check-list Scale (using printed version of specific self-administered questionnaires completed by the patient' close relative)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic PERENNOU, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; François RANNOU, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No